CLINICAL TRIAL: NCT03536351
Title: Building Social Skills With Interdisciplinary Drama With Children With Autism Spectrum Disorder
Brief Title: Building Social Skills With Interdisciplinary Process Drama in ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Lorie Richards, Chair and Associate Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB_0091961
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Autistic Disorder
Keywords: social skills; child; theory of mind; drama; occupational therapy; speech-language pathology; neural activation
MeSH Terms: conditions — Autistic Disorder; Social Skills

STUDY DESIGN:
Intervention Model Description: One group design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interdisciplinary process drama (Experimental): Process drama program (3 days/week, 12 weeks, 1-1.5 hours per session) of movement-based activities combining music and drama. Activities have been planned by a collaborative team of drama teachers, occupational therapists, and speech language pathologists, and target understanding emotion, intentions and appropriate social interactions.
  Interventions: Behavioral: Interdisciplinary process drama

INTERVENTIONS:
Behavioral: Interdisciplinary process drama — Process drama program (3 days/week, 12 weeks, 1-1.5 hours per session) of movement-based activities combining music and drama. Activities that target understanding of emotions, intentions, and appropriate social interactions have been planned by a team of drama teachers, occupational therapists, and speech-language pathologists.

SUMMARY:
This is a one group pre-post feasibility study of an interdisciplinary (theatre, Occupational Therapy (OT) and Speech Language Pathology (SLP)) intervention targeted at social skill development in children, aged 3-4. The intervention uses process drama modified with OT and SLP techniques and using typically developing peer models . Feasibility outcomes are recruitment rates, retention rates, daily program records of ease of implementing the program, and record of modifications needed. Child primary outcomes are Social Skills Improvement Scale (SSIS) and the Theory of Mind (ToM) Battery and Inventory within 4 weeks of program end. Secondary outcomes will be the Structured Play Assessment (SPA) within 4 weeks post-intervention, observations of social interactions (e.g.,eye contract, joint attention, verbal utterances, physical contact) during intervention sessions, brain activity in frontal and temporal/parietal areas during ToM tasks measured by high density EEG within 4 weeks of program end, and parental interview at 3 months related to child's social skills.

DETAILED DESCRIPTION:
Five children with Autism Spectrum Disorder (ASD) and 3-5 typically developing (TD) children will complete baseline testing. The TD children will only complete the EEG testing, while the ASD children and their parents will complete all outcome assessments. In addition to the outcome measures listed in the Brief Summary, we will administer the Vineland Adaptive Behavioral Scales (Vineland - II), the Mullen Scales of Early Learning, and the Autism Diagnostic Observation Scale - II (if they have not had one administered within the past 12 months) for sample description.

During the EEG session, brain activity during theory of mind and other social stimuli will be used to measure brain behavior relationships. The recordings will adhere to standard clinical EEG procedures, using high density EEG providing a high spatial resolution for electrical source imaging in brain space. They will be conducted by a Registered EEG Technologist (R. EEG T) with a specially trained student assistant. The procedure will involve first explaining to the parent and child what will be done. The participants will sit within a chair or a parent's lap while the EEG is recorded. The EEG tasks will consist of the following: First the child will be asked to open and close their eyes for a few minutes to record a baseline resting EEG. Then there will be both auditory sounds (intonations and word components) and images of social stimuli embedded between fun cartoon stimuli to maintain the child's attention displayed on a screen. The pictures will consist of eye movements, facial gestures, and point light diagrams of body movements.

The process drama program will be conducted with 5 children with ASD and 3-5 TD peer models 3 days per week for 12 week for 1-1.5 hours each day. The program will consist of several sections. Each day will open with an opening ritual that is movement based involving mirroring activity. This is followed by a welcome/greeting activity, involving things like a song and Name activity. The remainder of the activities build around a story for the day. The story will be one that holds interest for young children, such as a day in the life of a tree who gets visited by animals and people. The story unfolds with problems to solve and social interactions to do. Participants and the drama teachers take on different roles to bring out the story. Engagement starts out with drama pieces that the children can do individually and progress to those requiring a partner and then small groups. The sessions close with a closing ritual, reminding the participants of what was done during the session and a song. All the activities focus on building understanding the emotions and intentions of others and appropriate social interactions. The setting of the program and the specific activities have been planned with a collaborative team of drama teachers, an occupational therapists, and a speech language pathologists.

The process drama sessions will be taped and later scored for social interactions and social verbal and non-verbal communication. We will also examine the engagement of the participants with ASD to determine if we need to change/alter any procedures/techniques that we are using during the process drama sessions in subsequent versions of this research. We will also examine the behavior of the peer models to identify areas in which the research team may need to change to better engage the peer models in subsequent sessions.

After the end of the process drama intervention, the participants with ASD will repeat the baseline assessments within 4 weeks of intervention end. The assessments that will be repeated are the ToMT, SPA and SSiS. The children with ASD will also complete another EEG session as they did at baseline. Parents will be interviewed at 3 months post-intervention regarding changes in social skills.

ELIGIBILITY:
Inclusion Criteria: for children with ASD:

* aged 3-4 years old
* documented diagnosis of ASD from a licensed professional using DSM 5 criteria12; If no documentation available, meets cut off on Autism Diagnostic Observation Scale (ADOS -2)13 that will be administered by trained study staff.
* passes language and cognitive screen (see attached screening document with decision rules) and a receptive language age equivalence of ≥30 months and a non-verbal age equivalent score of ≥30 months on the Mullen Scale of Early Learning
* have a caregiver willing/able to bring them to the University for the study sessions and to schedule up to 3 assessment visits prior to intervention start and 3 assessment sessions after intervention end
* family's primary language is English

INCLUSION for TD children:

* aged 3-4
* normal or corrected to normal vision and hearing
* English speaking

Exclusion Criteria: for children with ASD:

* have no other major medical conditions (i.e., no genetic disorders such as Fragile X, Down syndrome)
* seizure disorder
* uncorrected hearing or visual impairment
* other condition causing motor impairment, such as Cerebral Palsy

Exclusion for TD children:

* history of developmental delay or neurological disorder

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Social Skills Improvement Scale | 4 weeks post intervention
  Parent rating of statements about child's social interactions as never, seldom, often, almost always. These are transformed to numeric scores, varying with the content of the item, either ranging from 0-3 or 1-3. Each subscale has a different number of items. Subscales of communication, cooperation, assertion, responsibility, empathy, engagement, self-control scores, externalizing problem behaviors, bullying, hyperactivity/inattention, and internalizing problem behaviors items are summed to obtain subscale raw scores, which are translated into "below average", "average", and "above average", based on age and gender normative data. The autism spectrum subscale is scored the same way.
Theory of Mind Battery & Inventory | 4 weeks post intervention
  Performance test of ToM activities and parent ratings of statements of child behavior in ToM situations
recruitment | pre intervention
  ability to recruit needed number of participants in time frame availability
retention | 4 weeks post- and 3 months post-intervention
  number of participants who completed 4 week assessment and parental interview

SECONDARY OUTCOMES:
Structured Play Assessment | 4 weeks post intervention
  performance test of how child plays with toys
Brain activity during ToM tasks | 4 weeks post intervention
  Dense EEG recordings of brain activity in front/temporal/parietal areas during ToM tasks
Parental perceptions of social skills | 3 months post intervention
  interview with parent regarding changes seen in social skills
Changes in social skills during program | 12 weeks during program
  observations (via digital recordings) of social skills during intervention program
modifications needed to program | 12 weeks during program
  record of modifications to the program during the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lorie G Richards, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Corbett BA, Key AP, Qualls L, Fecteau S, Newsom C, Coke C, Yoder P. Improvement in Social Competence Using a Randomized Trial of a Theatre Intervention for Children with Autism Spectrum Disorder. J Autism Dev Disord. 2016 Feb;46(2):658-72. doi: 10.1007/s10803-015-2600-9. PMID 26419766
- [Result] Pelphrey KA, Morris JP, McCarthy G. Grasping the intentions of others: the perceived intentionality of an action influences activity in the superior temporal sulcus during social perception. J Cogn Neurosci. 2004 Dec;16(10):1706-16. doi: 10.1162/0898929042947900. PMID 15701223
- [Result] Thomas MS, Davis R, Karmiloff-Smith A, Knowland VC, Charman T. The over-pruning hypothesis of autism. Dev Sci. 2016 Mar;19(2):284-305. doi: 10.1111/desc.12303. Epub 2015 Apr 6. PMID 25845529